CLINICAL TRIAL: NCT04576299
Title: Health Care Workers' Perception of Patient Safety During the COVID-19 Pandemic: Opportunities and Challenges
Brief Title: Health Care Workers' Perception of Patient Safety During COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Universidad de Santander (Other); Universidad Antonio Nariño (Other); University of Sao Paulo (Other); Universidad Catolica Santiago de Guayaquil (Other); Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, José Joaquín Mira, Professor, Universidad Miguel Hernandez de Elche
Other Study IDs: 2020-09
Record Dates: First submitted 2020-09-28; First posted 2020-10-06 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Patient Safety
Keywords: Patient Safety; Healthcare Personnel; Hospital Management

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthcare workers.: Survey developed specifically for the objective of this study: Healthcare worker perception of patient safety in times of pandemic.
  The application will be done through a digital questionnaire in the surveymonkey platform (Link of the instrument: https://es.surveymonkey.com/r/COVIDSP)
  Interventions: Other: Group 1

INTERVENTIONS:
Other: Group 1 — Survey about social networks, notification of adverse events, multidisciplinary teams, the doctor-patient relationship, the role of the ethics and patient safety committees, protocol compliance and suspension of outpatient procedures
  Other Names: COVID-PS HW

SUMMARY:
Objective: Analyze health care workers' perception of patient safety during the COVID 19 pandemic.

Methodology: Analytical cross-sectional observational study, with a quantitative focus on healthcare workers who are working on-site during the pandemic in the services of healthcare institutions that agree to participate in the countries where the study will be conducted, by applying a survey of patient safety perceptions in healthcare workers in times of pandemic. Analysis of the data will employ descriptive and inferential statistical techniques to meet the objectives of the study using IBM SPSS Statistics for Windows version 25.0 software.

Expected results: The study seeks to generate evidence for the perception of patient safety in times of pandemic, for which it will generate the submission of an article with the results obtained to an indexed journal and presentation at a scientific event.

DETAILED DESCRIPTION:
Introduction

Patient safety culture The concept of patient safety culture has become one of the strategies in health care institutions that seeks to intervene on adverse events, understood as: the set of characteristics, skills and attitudes, perceptions, abilities, competencies, among others, that are developed within the institutions and their members, which establish the commitment and capabilities to maintain and manage safety in health care in all processes that are developed within the organization. The issue of safety culture is part of the DNA of each organization, involving their operational processes and the perspective of how they manage them, with a view to becoming "highly reliable organizations", being institutions that despite working in very high risk situations, the presence of adverse events, accidents or complications is very low.

Therefore, it is important to understand the patient's perception of safety that allows the evaluation of dimensions such as: commitment of the directives, processes of institutional continuous improvement, systems of notification of events and incidents, communication and climate of confidence, fundamental dimensions at the moment of measuring the culture. However, it is also important to assess how these dimensions have been impacted at times of a pandemic such as the current COVID19 , where around 29,000,000 positive cases and 1 million deaths are reported worldwide, a situation for which institutions and countries were not prepared and which may impact on patient safety processes, mediated by high levels of stress and anxiety in the health team work overload due to increased care and disability leave of workers who have acquired the virus.

Therefore, this study seeks to examine health care workers' perceptions of patient safety during the COVID 19 pandemic.

Rationale

Given the environmental, social and economic impacts that the current SARS-CoV-2 pandemic is having on all population dynamics, it is important to highlight the effects it is having on the health sector, since it is there that it is directly involved in the access, treatment, control and resolution of patients with this pathology. Precisely its human capital, where health professionals are located, is the most representative and numerous population in the various processes and actions carried out within it. The positive or negative results related to the management of SARS-CoV-2 in users depend on this personnel.

From the aspects highlighted by the World Health Organization and the Pan American Health Organization, given the situation of direct exposure to the virus through contact with health teams and its high increase in infections and deaths of health personnel, agree to promote protection strategies such as establishing standard procedures for prevention and control of infections, increase in the number of personal protective equipment (PPE), expansion in the processes of retraining, flexible workloads and increased staff.

Although there are various initiatives and interventions by health institutions and national governments in response to this situation of security for health personnel, concern is further increased by the increase in the number of Covid - 19 infections, by August 2020 in the epidemiological alert of the Americas for this situation in health personnel, the panorama is as follows. The most affected countries are Brazil, Mexico, Argentina and Colombia.

On the Brazilian side, with a total of 268,954 confirmed cases in their health team, the nursing auxiliaries and nurses are the most impacted with 34% and 14% of these cases respectively. On the other hand, in Mexico the confirmed cases in the health personnel ascends to 97,632 people, the professional nursing is the most impacted work with 42% of the total of the professionals.

In third place in Latin American, Argentina has reported a total of 16,194 cases among young people between the ages of 29 and 39. In the case of Colombia, there are currently 7,692 cases, with a greater proportion of nurses and doctors.

According to the above, this research seeks to analyze the perception of patient safety of health workers in Latin American countries during the COVID 19 pandemic. Due to the deficit of knowledge and the situation related to the impacts on health professionals, in the same way few initiatives deepen the generation of knowledge about this problem at the local level, this work is convenient to consolidate more effective actions in view of the increase of cases of health personnel.

On the other hand, the research contributes to expand the linkage of patient safety in health organizations, the work of the professional and the improvement of processes according to the realities that are presented in each of the services, units, institutions that are adapting to the changing situations and variables of the pandemic.

The work has a methodological utility since future research could be carried out related to the subject of hospitals or health institutions at different levels of care, the permanent training of human capital and the improvement of processes according to the adaptations in the management of the care units.

Problem Statement

The culture of patient safety has become the main strategy to mitigate and manage the presentation of adverse events related to health care. Faced with this phenomenon, studies have been carried out related to the validation of instruments that allow measuring the perception of workers and members of the health teams of the institutions of each of the dimensions of the organizational culture associated with safety, which they measure from the commitment of senior management, as communication strategies of the adverse event, job satisfaction, rewards and recognition, teamwork, working conditions, individual factors, attitudes and practices, continuous improvement process, among others, that have used construction validations, internal consistency and viability presenting very good results. Among these reported instruments are: safety attitudes questionnaire (SAQ), Veteran Affairs Palo Alto/Stanford Patient Safety Center for Inquiry PSCI =Patient Safety Climate in Healthcare Organizations PSCHO, AHRQ Hospital Survey on Patient Safety Culture, Safety Climate Survey, modified ORMAQ and Safety Climate Scale, among others.

To this extent, research has shown the following to be fundamental factors in the patient safety culture: the participation of management and process leaders as indispensable elements for the promotion and prioritization of patient safety issues, and where studies report low commitment and interest at this level, the use of anonymous event reporting systems and with the use of information and communication technologies, as well as low coordination and teamwork among units and members of the same team that is also perceived as leadership failures.

Therefore, it is clear that there are great advances in measuring the culture of safety in health institutions, but this measurement has not been carried out in situations where health systems worldwide are collapsed and have great difficulties in responding to a pandemic, as is currently the case with COVID 19, where intensive care and emergency services have reached occupations of over 90%, which implies a greater work overload, and can interfere negatively with the safe attention to users, also given by high levels of stress and anxiety in the health team that has been shown to be related to aspects to be improved around this problem in previous studies, and which make the presentation of errors and incidents in health care more likely. Thus, this study seeks to analyze the perception of patient safety in the members of the health team during this pandemic, allowing the generation of evidence that will enable health systems and institutions to take action on the findings of the study and to strengthen, if necessary, those dimensions with negative perceptions that will allow a better response to this situation.

Research question:

What is the patient safety perception of health workers during the COVID 19 pandemic in 2020?

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professionals from all disciplines
* Technicians from all disciplines (health related)
* Working in a face-to-face manner during the pandemic in the services of health institutions
* Professional or technical personnel in charge of the quality and patient safety processes in the institutions.

Exclusion Criteria:

* Professional or technical staff from the administrative areas

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthcare workers and patient safety coordinators from the participant countries (Brazil, Chile, Colombia, Ecuador).
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Patient Safety perception. | 30 days
  Differences of patient safety perceptions among the participants from different countries.
  An ad-hoc survey questionnaire (not validated) has been developed by researchers using prior tools and personal experience by means of virtual conference consensus. The survey includes 32 questions about social networks, notification of adverse events, multidisciplinary teams, the doctor-patient relationship, the role of the ethics and patient safety committees, protocol compliance and suspension of outpatient procedures using a likert scale of 5 possible answers (totally disagree - totally agree).

CONTACTS AND LOCATIONS:
Overall Officials: Jose J Mira, PhD, Principal Investigator — Professor
Locations (4):
- Pontificia Universidad Católica de Chile, Santiago, Chile
- Universidad de Santander, Bucaramanga, Santander Department, Colombia
- Universidad Católica de Santiago de Guayaquil, Guayaquil, Guayas, Ecuador
- Miguel Hernández University, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Antino, M., Sanchez-Manzanares, M., & Ortega, A. (2020). The hospital survey on patient safety culture in Mexican hospitals: Assessment of psychometric properties. Safety Science, 128(May 2017), 104706. https://doi.org/10.1016/j.ssci.2020.104706
- [Background] Arias-Botero, J. H., & Gómez-Arias, R. D. (2017). La cultura de la seguridad del paciente: enfoques y metodologías para su medición. Ces Medicina, 31(2), 180-191. https://doi.org/10.21615/cesmedicina.31.2.7
- [Background] Camargo Tobias, G., Queiroz Bezerra, A. L., & Silvestre Branquinho, N. C. (2014). Cultura de la seguridad del paciente en la atención sanitaria: Un estudio bibliométrico. Enfermeria Global, 13(1), 336-361. https://doi.org/10.6018/eglobal.13.1.159931
- [Background] Huang L, Lei W, Xu F, Liu H, Yu L. Emotional responses and coping strategies in nurses and nursing students during Covid-19 outbreak: A comparative study. PLoS One. 2020 Aug 7;15(8):e0237303. doi: 10.1371/journal.pone.0237303. eCollection 2020. PMID 32764825
- [Background] Pinheiro da Penha, M., Junior da Silva, O., da Penha Pinheiro, M., & da Silva Júnior, O. (2017). Evaluación de la cultura de seguridad del paciente en una organización hospitalaria de un hospital universitario. Enfermería Global: Revista Electrónica Semestral de Enfermería, 16(1), 309-352.
- [Background] Ramos, F., Coca, S. M., & Abeldaño, R. A. (2017). Percepción de la cultura de seguridad de pacientes en profesionales de una institución argentina. Enfermería Universitaria, 14(1), 47-53. https://doi.org/10.1016/j.reu.2016.12.004
- [Background] Singer S, Meterko M, Baker L, Gaba D, Falwell A, Rosen A. Workforce perceptions of hospital safety culture: development and validation of the patient safety climate in healthcare organizations survey. Health Serv Res. 2007 Oct;42(5):1999-2021. doi: 10.1111/j.1475-6773.2007.00706.x. PMID 17850530
- [Background] University Johns Hopkins. (2020). COVID-19 Dashboard by the Center for Systems Science and Engineering (CSSE) at Johns Hopkins University (JHU). https://gisanddata.maps.arcgis.com/apps/opsdashboard/index.html#/bda7594740fd40299423467b48e9ecf6
- [Background] Zhu Z, Xu S, Wang H, Liu Z, Wu J, Li G, Miao J, Zhang C, Yang Y, Sun W, Zhu S, Fan Y, Chen Y, Hu J, Liu J, Wang W. COVID-19 in Wuhan: Sociodemographic characteristics and hospital support measures associated with the immediate psychological impact on healthcare workers. EClinicalMedicine. 2020 Jun 24;24:100443. doi: 10.1016/j.eclinm.2020.100443. eCollection 2020 Jul. PMID 32766545
- See also: Be+ Against COVID Second Victims working group website — https://secondvictimscovid19.umh.es/p/home.html